CLINICAL TRIAL: NCT01904045
Title: A Multicentre, Prospective, Non-Interventional Study to Assess the Intra-patient Variability of Tacrolimus Once and Twice Daily After Kidney Transplantation
Brief Title: PEL-1235_REN-0176-I (Pelicon)
Acronym: Pelicon
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: PEL-1235_REN-0176-I
Record Dates: First submitted 2013-07-02; First posted 2013-07-22 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Immunosuppression After Kidney Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Other: tacrolimus Advagraf — intake of Advagraf once daily for 3 months
Other: tacrolimus Prograf — intake of Prograf twice daily for 3 months

SUMMARY:
Aim of this study is to investigate whether in patients following kidney transplantation (>6 months after transplantation), the intra-patient variability of levels of tacrolimus is comparable after administration of tacrolimus twice daily (Prograf) to tacrolimus once daily (Advagraf), with each regimen for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* male or female patient ≥ 18years of age
* Patient has received a kidney transplantation at least 6 months prior to inclusion into the study
* No acute rejection episodes for at least 3 months
* PRG through level and dosing stable for at least 1 month
* Patient is capable of understanding the purpose and risks of the study, has been fully informed and has given written informed consent to participate in the study

Exclusion Criteria:

* Acute rejection episodes within the last 3 months prior to study entry
* Unstable PRG trough level or dose change in the month before study entry
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Treatment with another investigational product during this study or during the last 30 days prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2018-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Intrapatient variability of tacrolimus through level | pre-dose, 1 h post dose and 3 h post dose for 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, Department of Nephrology, Munich, Bavaria, Germany